CLINICAL TRIAL: NCT03178110
Title: Effectiveness of Manual Therapy in Combination With a Dynamic Splint (Dynasplint) in the Treatment of Trismus in Patients With Head and Neck Cancer: A Pilot Study
Brief Title: Manual Therapy and Use of the Dynasplint for Trismus in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREBA-CC-17-0164
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Neoplasms, Head and Neck; Trismus
Keywords: physical therapy; cancer rehabilitation
MeSH Terms: conditions — Head and Neck Neoplasms; Trismus | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: The methodology of a single subject design will be used with multiple baseline and during treatment measures to determine the effectiveness of the treatment protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical therapy and dynasplint (Experimental): Participants with trismus will receive a manual therapy protocol plus exercises and the use of the dynasplint (DTS) device for a duration of 8 weeks. The first two weeks of treatment will include 2 days per week of manual therapy and active jaw opening exercises. Following this initial treatment phase, the DTS will be introduced and the frequency of manual therapy will remain at two times per week.
  Interventions: Behavioral: Physical therapy and dynasplint

INTERVENTIONS:
Behavioral: Physical therapy and dynasplint — Participants will receive a session of 30-45 minutes of manual therapy two times per week, for eight weeks. All participants will be instructed how to use the Dynasplint® Trismus System at home. Participants will start the use of the DTS for 10-30 minutes three times per day, every day. If the exercises are well tolerated, time will be progressively increased to 30 minutes and then intensity (force) will be increased.

SUMMARY:
The objectives of this pilot study are to determine the effectiveness of a manual therapy (MT) protocol plus the use of a dynamic jaw opening device on the maximal interincisor distance; on trismus symptoms; on pain-disability outcomes and on the quality of life, anxiety, and depression in subjects with trismus. The proposed pilot study will comprise a single subject design with multiple baseline measures and during treatment phases to determine the effectiveness of the treatment protocol. A minimum sample of 10 subjects will be recruited. The Health Research Ethics Board of Alberta Cancer Committee will approve this study. Participants will receive a MT protocol plus exercises and the use of the DTS device for 8 weeks. The first two weeks of treatment will involve only MT and opening exercises.After this initial 2 weeks, the DTS will be introduced. The participants will receive a session of 30-45 minutes of MT three/two times per week, for 8 weeks. All participants will be instructed how to use the Dynasplint® Trismus System at home.

Analyses: Visual analyses will be performed on participant before, during, and after the intervention. The 2-standard deviation band method will be used to analyze the behavior of each participant on the outcome of interest before, during, and after the treatment. The minimally important difference levels in order to determine clinical relevance will be done. Two effect size indexes will be used: the percentage of non-overlapping data, and the percentage of improvement rate difference.

DETAILED DESCRIPTION:
Trismus is a common impairment following treatment for head and neck cancer. The prevalence of trismus ranges from 25% to 46%, and may be the result of a tumour growth, infection, surgery or radiation. Trismus can dramatically affect the quality of life of subjects with cancer in a variety of ways, and may contribute to post treatment depression. Early intervention is key to reduce the chances of complications. Multiple modalities have been used in the treatment of trismus: Physical therapy, hyperbaric oxygen and pentoxifylline, forced mouth opening under general anesthesia, surgical coronoidectomy, botulinum toxin injection and jaw opening devices such as the TheraBite Jaw Motion Rehabilitation and the Dynasplint® Trismus System. Manual therapy (MT) constitutes a wide variety of different techniques which may be categorized into four major groups: manipulation, mobilization, and muscle energy techniques. MT in the form of mobilization associated with exercises has been frequently used to treat temporomandibular disorders (TMD) with promising results. The Dynasplint® Trismus System (DTS) is a jaw opening device used as a self-management strategy for trismus. The DTS provides low-torque, prolonged-duration stretching with the aim of lengthening the affected connective tissue permanently.Positive effects of the use of DTS in patients with trismus to increase mouth opening have been reported. To date, however, the evidence is limited regarding the effectiveness of manual therapy alone or in combination with exercises to treat specifically trismus in patients with head and neck cancer.

The main objectives of this project are: 1) To determine the feasibility and preliminary efficacy of a manual therapy protocol plus the use of a dynamic jaw opening device (DTS) on the maximal interincisor distance (MID) in subjects with trismus.

2) To determine the preliminary efficacy the manual therapy protocol plus the use of a dynamic jaw opening device (DTS) on the Gothenburg Trismus Questionnaire (GTQ). 3) To determine the preliminary efficacy of a manual therapy protocol plus the use of a dynamic jaw opening device (DTS) on pain-disability outcomes in subjects with trismus.

4) To determine the preliminary efficacy of a manual therapy protocol plus the use of a dynamic jaw opening device (DTS) on the quality of life, anxiety, and depression in subjects with trismus.

This study will be a pilot study and will follow the methodology of a single subject design with multiple baseline measures and during treatment phases to determine the effectiveness of the treatment protocol. The single subject design was chosen because in addition to provide sound research results, clinical significance of the results for a specific group of patients can be derived. Thus, variables that are functionally important for treatment can become evident. The multiple baseline measures will be used because it increases the potential number of comparisons that can be made between and within data series, ultimately strengthening the confidence with which conclusions are made from the data. A minimum sample of 10 subjects who attend the Cross Cancer Institute (CCI) in Edmonton will be recruited for this project. Subjects will be screened for eligibility and if they meet all eligibility criteria, an information letter of the study will be provided and they will be asked to sign a consent form according to the Health Research Ethics Board (HREB) - University of Alberta.

Participants with trismus will receive a manual therapy protocol plus exercises and the use of the DTS device for a duration of 8 weeks twice per week. The first two weeks of treatment, treatment will involve only manual therapy and opening exercises. After this initial 2 weeks, the DTS will be introduced.

Physical Therapy: The participants will receive a session of 30-45 minutes of manual therapy three/two times per week, for eight weeks. Every sessions will be done and will be adapted individually to the needs of each subject.

Home Exercises: All participants will be instructed how to use the Dynasplint® Trismus System (DTS; Dynasplint Systems Inc, Severna Park, Md, USA) at home. Participants' initial introduction to the DTS will include customized fitting (molded patient mouth pieces) and training on donning and doffing of the devices. Verbal and written instructions will be provided throughout the duration of the treatment for safety, general wear and care, and tension setting goals, based on patient tolerance. Participants will start the use of the DTS for 10-30 minutes three times per day, every day. If the exercises are well tolerated, the tension will be increased every 2 weeks until maximum tolerance is reached. Participants will use this device for the duration of the manual therapy and exercise protocol.

Statistical Analysis: To analyse the data, visual analyses will be done. This kind of analyses is really important for single subject design research to determine: whether evidence of a relation between an independent variable and an outcome variable exists and the strength or the magnitude of that relation. The visual analyses will show the behavior of each participant before, during, and after the intervention. The 2-standard deviation band method (2-SD) will be used to analyze the behavior of each participant on the outcome of interest before, during, and after the treatment. Two effect size indexes will be used to analyse the data. The first one will be the percentage of non-overlapping data (PND), that is obtained by counting the number of data points in the intervention phase which do not overlap with the highest or lowest data points in the baseline phase; this number then is divided by the total number of data points in the treatment phase, multiplied by 100. The second effect size index will be the percentage of improvement rate difference (IRD), that considers the difference in successful performance between baseline and intervention phases. The main purpose of using these two effect sizes is to explore the effects of treatment and to describe the phase contrast and design context.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of head and neck cancer;
2. Cancer treatment includes surgery and/ or radiation therapy;
3. An oral and an opening of less than 35 mm between the upper and lower incisors (measured with a slide caliper).

Exclusion Criteria:

1. 17 years or younger;
2. Osteoporosis, osteoradionecrosis or active cancer in the region;
3. Serious or uncontrolled co-morbid disease that would interfere with testing or treatment;
4. Inability to provide informed consent;
5. Inability to comply with the assessment and/ or treatment (i.e. unable to attend treatment sessions due to vacation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Minimal Inter-incisor Opening | 8 weeks
  Mouth Opening

SECONDARY OUTCOMES:
Gothenburg Trismus Questionnaire | 8 weeks
  Trismus symptoms
Visual Analogue Scale for Pain | 8 weeks
  10 cm scale for pain
Hospital Anxiety and Depression Scale | 8 weeks
  Brief psychological screening instrument to measure psychological distress
Short-Form 36 Health Survey | 8 weeks
  SF-36 health-related quality of life questionnaire
Global Rating Scale | 8 weeks
  Scale to assess the magnitude of change experienced in pain and jaw function
Adherence to protocol | 8 weeks
  Diary of adherence to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Margaret McNeely, PhD, Principal Investigator — University of Alberta; Susan Olivo, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta/ Cross Cancer Institute, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Undecided
No plan in place at this time.